CLINICAL TRIAL: NCT01697878
Title: Consequences of Obstructive Sleep Apnea on Respiratory Function Following Weight-loss Surgery: A Randomized Controlled Trial
Brief Title: Consequences of Obstructive Sleep Apnea on Respiratory Function Following Weight-loss Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Matthias Eikermann, Assistant Pofessor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011P001333; ResMed (Other Grant/Funding Number: 2011D001139)
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Obstructive Sleep Apnea; Obesity
Keywords: obstructive sleep apnea; obesity; respiratory function; weight loss surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomization Group 1 (Experimental): CPAP first followed by standard of care
  Interventions: Procedure: CPAP followed by atmospheric pressure
- Randomization group 2 (Active Comparator): Standard of care followed by CPAP
  Interventions: Procedure: Atmospheric pressure followed by CPAP

INTERVENTIONS:
Procedure: CPAP followed by atmospheric pressure — In the PACU, Patients receive 2 hours of continuous-positive-airway-pressure (CPAP) oxygen at 30% FiO2 treatment followed by 2 hours of oxygen treatment (6 L O2/min) that is part of standard of care at Massachusetts General Hospital
  Other Names: Tx Plan 1
  Arms: Randomization Group 1
Procedure: Atmospheric pressure followed by CPAP — In the PACU, patients receive 2 hours of Oxygen treatment (6L/min) that is part of standard-of-care at Massachusetts General Hospital, followed by 2 hours of Continuous Positive Airway Pressure (CPAP) treatment at 30% FiO2.
  Other Names: Tx Plan 2
  Arms: Randomization group 2

SUMMARY:
The investigators propose to compare two different treatments, continuous positive airway pressure (CPAP) versus breathing of atmospheric pressure, in subjects with obstructive sleep apnea (OSA)recovering from weight loss surgery in the post anesthesia care unit (PACU). WE hypothesize that subjects with OSA will have a higher Apnea-Hypopnea Index (AHI) with desaturation and the investigators expect that post-operative CPAP treatment in the PACU will significantly improve the AHI and therefore improve patient safety in the PACU. The investigators also hypothesize that subjects with OSA have a greater decrease in oxygen saturation in response to opioid administration by patient-controlled opioid analgesia (PCA).

DETAILED DESCRIPTION:
Patients with morbid obesity have an approximately 60-80 percent incidence of OSA depending on the criteria used for making diagnosis, and they are suggested to be at increased risk to develop serious perioperative complications, especially during the postoperative period. Weight loss might be considered as an appropriate treatment of OSA but in turn it has recently been reported that OSA is an independent risk factor for development of perioperative complications, importantly oxygen desaturation, in patients undergoing weight loss surgery. It seems logical to evaluate if these patients would benefit from post-operative CPAP treatment in the PACU. The results of this multidisciplinary study will have an impact on PACU treatment of patients with OSA and will further optimize patient care at MGH.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for weight loss surgery at Massachusetts General Hospital
* Male and female subjects
* age ≥ 18 years

Exclusion Criteria:

* CNS disease with impairment of cognitive function and/or muscle paresis such as stroke, or dementia
* age < 18 years
* missing or insufficient PSG data to make diagnosis OSA
* impaired decision making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
apnea hypopnea index (AHI) | preoperatively for one night of sleep and during 2 hours of recovery room stay
  The AHI is assessed for one night's sleep in the initial at-home sleep study conducted with a portable Alice monitor. Subsequently, the AHI is assessed during the patient's stay in the post-anesthesia-care unit (PACU) during which time they receive CPAP and oxygen treatment.

SECONDARY OUTCOMES:
apneas after opioid bolus self-administration | 5 minutes after each opioid PCA administration
  We are assessing the effects of OSA on apneas occurring in a 5 minute time-frame after opioid bolus self administration in the PACU, and consider these as related to opioid administration

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD-PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Malbois M, Giusti V, Suter M, Pellaton C, Vodoz JF, Heinzer R. Oximetry alone versus portable polygraphy for sleep apnea screening before bariatric surgery. Obes Surg. 2010 Mar;20(3):326-31. doi: 10.1007/s11695-009-0055-9. Epub 2010 Jan 6. PMID 20052560
- [Background] Longitudinal Assessment of Bariatric Surgery (LABS) Consortium; Flum DR, Belle SH, King WC, Wahed AS, Berk P, Chapman W, Pories W, Courcoulas A, McCloskey C, Mitchell J, Patterson E, Pomp A, Staten MA, Yanovski SZ, Thirlby R, Wolfe B. Perioperative safety in the longitudinal assessment of bariatric surgery. N Engl J Med. 2009 Jul 30;361(5):445-54. doi: 10.1056/NEJMoa0901836. PMID 19641201
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Faccenda JF, Mackay TW, Boon NA, Douglas NJ. Randomized placebo-controlled trial of continuous positive airway pressure on blood pressure in the sleep apnea-hypopnea syndrome. Am J Respir Crit Care Med. 2001 Feb;163(2):344-8. doi: 10.1164/ajrccm.163.2.2005037. PMID 11179104
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Meoli AL, Rosen CL, Kristo D, Kohrman M, Gooneratne N, Aguillard RN, Fayle R, Troell R, Kramer R, Casey KR, Coleman J Jr; Clinical Practice Review Committee; American Academy of Sleep Medicine. Upper airway management of the adult patient with obstructive sleep apnea in the perioperative period--avoiding complications. Sleep. 2003 Dec 15;26(8):1060-5. doi: 10.1093/sleep/26.8.1060. PMID 14746392
- [Background] Loadsman JA, Hillman DR. Anaesthesia and sleep apnoea. Br J Anaesth. 2001 Feb;86(2):254-66. doi: 10.1093/bja/86.2.254. PMID 11573670
- [Background] Hillman DR, Loadsman JA, Platt PR, Eastwood PR. Obstructive sleep apnoea and anaesthesia. Sleep Med Rev. 2004 Dec;8(6):459-71. doi: 10.1016/j.smrv.2004.07.002. PMID 15556378
- [Background] Mezzanotte WS, Tangel DJ, White DP. Influence of sleep onset on upper-airway muscle activity in apnea patients versus normal controls. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1880-7. doi: 10.1164/ajrccm.153.6.8665050.
- [Background] Hajiha M, DuBord MA, Liu H, Horner RL. Opioid receptor mechanisms at the hypoglossal motor pool and effects on tongue muscle activity in vivo. J Physiol. 2009 Jun 1;587(Pt 11):2677-92. doi: 10.1113/jphysiol.2009.171678. Epub 2009 Apr 29. PMID 19403616
- [Background] White DP. Opioid-induced suppression of genioglossal muscle activity: is it clinically important? J Physiol. 2009 Jul 15;587(Pt 14):3421-2. doi: 10.1113/jphysiol.2009.176388. No abstract available. PMID 19602634
- [Background] Gross JB, Bachenberg KL, Benumof JL, Caplan RA, Connis RT, Cote CJ, Nickinovich DG, Prachand V, Ward DS, Weaver EM, Ydens L, Yu S; American Society of Anesthesiologists Task Force on Perioperative Management. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: a report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2006 May;104(5):1081-93; quiz 1117-8. doi: 10.1097/00000542-200605000-00026. No abstract available. PMID 16645462